CLINICAL TRIAL: NCT02439736
Title: A PROSPECTIVE CLINICAL EVALUATION OF BIOMARKERS OF TRAUMATIC BRAIN INJURY EXTENSION STUDY
Brief Title: EVALUATION OF BIOMARKERS OF TRAUMATIC BRAIN INJURY EXTENSION STUDY
Acronym: ALERT-TBIx
Status: Completed | Type: Observational
Sponsor: Banyan Biomarkers, Inc (Industry)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: ATO-06x
Record Dates: First submitted 2015-05-07; First posted 2015-05-12 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Head Injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CT positive for acute intracranial lesion
  Interventions: Other: Blood draw within 12 hours of head injury

INTERVENTIONS:
Other: Blood draw within 12 hours of head injury

SUMMARY:
The primary objective of this study is to evaluate Ubiquitin C-terminal Hydrolase-L1 (UCH-L1) and Glial Fibrillary Acidic Protein (GFAP) biomarker levels in a population of CT-positive subjects (as determined by an independent Neuroimaging Review Committee) presenting acutely with traumatic brain injury (Glasgow Coma Scale score 9-15).

ELIGIBILITY:
Inclusion Criteria:

* The Subject is at least 18 years of age at screening.
* The Subject has presented to a Health Care Facility (HCF) or Emergency Department (ED) with a suspected traumatically induced head injury, as a result of insult to the head from an external force.
* A Glasgow Coma Scale score of 9-15 at the time of Informed Consent.
* The subject is CT-positive for acute intracranial lesion(s) based on the local neuroradiologist's review of the subject's head CT scan.
* The CT scan and CT report used to determine eligibility must be available.
* The blood sample is collected as close to the time of head injury as possible, but no later than 12 hours.
* The Subject or their legal representative is willing to undergo the Informed Consent process prior to enrollment into this study

Exclusion Criteria:

* Participating in an interventional, therapeutic clinical study that may affect the results of this study (an observational study would be acceptable).
* Time of injury cannot be determined.
* Primary diagnosis of ischemic or hemorrhagic stroke.
* Venipuncture not feasible (i.e., skin integrity compromised at the venipuncture sites, blood vessel calcification (i.e., IV drug users, advanced atherosclerosis) both upper limbs missing (congenital or amputee)).
* The subject has a neurodegenerative disease or other neurological disorder including dementia, Parkinson's disease, multiple sclerosis, seizure disorder, or brain tumors.
* The subject has a history of neurosurgery within the last 30 days.
* Administration of blood transfusion after head injury and prior to the study blood draw.
* The subject is a female who is pregnant or lactating.
* The Subject is otherwise determined by the Investigator to be an unsuitable candidate for participation. If this criterion applies, a reason must be provided

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects eligible for study participation will be over the age of 18 with a standard of care head CT that has been confirmed to be CT-positive for acute intracranial lesions based on the local neuroradiologist's review and can undergo blood draw within 12 hours of head injury. Subjects who will be permitted into the study include those who will meet all the inclusion criteria and will have none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2015-06; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Correlation of assay results with presence of acute intracranial lesions | Day 1

CONTACTS AND LOCATIONS:
Locations (7):
- United States (5):
  - University of California San Diego, San Diego, California
  - Wayne State University - Detroit Receiving Hospital, Detroit, Michigan
  - Baylor College of Medicine/Ben Taub General Hospital, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
- Germany (2):
  - Ludwig-Maximilians-University, Munich
  - Klinikum rechts der Isar of the Technical University of Munich, Munich